CLINICAL TRIAL: NCT00660465
Title: Exploring the Relationship Between Varying CO2 Levels and the Regional BOLD Signal, by Using Breathing Exercises .
Brief Title: Exploring the Relationship Between Varying CO2 Levels and the Regional BOLD Signal, by Using Breathing Exercises
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Alexander Gersten, Ben-Gurion University of the Negev
Other Study IDs: SOR467608CTIL
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Regional BOLD signal dependency on arterial PaCO2.; Effect of breathing exercises on brain regional O2 level.; Healthy subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A18

SUMMARY:
The purpose of this study is to explore how arterial PaCO2 effect regional Blood Oxygen Level Dependent (BOLD) signal, and indirectly the brain regional O2 level .

DETAILED DESCRIPTION:
Among many parameters effecting cerebral blood flow(CBF), partial pressure of CO2 (PaCO2) in arterial blood has a significant effect. A small increase in arterial PaCO2 level will cause a significant increase of CBF , followed by increase of O2 level . The main objective is to explore the effect of arterial PaCO2 level on regional CBF and brain O2 level, by using breathing exercises to modulate arterial PaCO2. The regional Blood Oxygen Level Dependent (BOLD) signal produced by MRI , will indicate the regional O2 level.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years old .

Exclusion Criteria:

* under 18 years old.
* Artificial pacemaker
* implantable cardioverter-defibrillator (ICD)
* Hearing aid, implantable or portable.
* artificial heart valve
* Surgical clips
* Metal fragments in eyes
* Electronic stimulators
* Implanted pumps
* Implantable Neurostimulation Device
* metal fragments of any sort
* Permanent makeup or tattoo
* transfusion pump
* pregnant or breast feeding women
* False teeth , retainer or dental crown

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Shelef, M.D, Study Director — Head, Neuroradiolgy Unit ;Department of Diagnostic Imaging ;Soroka Univrsity Medical Center
Locations (1):
- Department of Diagnostic Imaging ;Soroka Univrsity Medical Center, Beersheba, Israel